CLINICAL TRIAL: NCT06270095
Title: " Évènements Feux/Fumées/Odeurs Lors Des Vols aériens : conséquences Sur la qualité de l'Air à l'intérieur Des Cabines d'Avions et Sur la santé Des Personnels Navigants d'Une Flotte aérienne française " (AviSan)
Brief Title: " Fume Events in Air Flights: Consequences on Cabin Air Quality and on Aircrews Health of a French Fleet of Aircraft"
Acronym: AVISAN
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Université Paris Cité (Other); National Agency for Sanitary Safety of the Food of the Environment and Labor (Other Government)
Responsible Party: Sponsor
Other Study IDs: C21-57
Record Dates: First submitted 2023-12-27; First posted 2024-02-21 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Neurologic Symptoms; Neurologic Disorder
Keywords: Fume events; Aircrew; Air quality; Organophosphorus compounds; Occupational exposure
MeSH Terms: conditions — Neurologic Manifestations; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Aircrew exposed to a fume event
  Interventions: Diagnostic Test: Neurocognitive, neuromuscular and neurosensitive tests.
- Non-exposed: Aircrew not exposed to a fume event but present on a control flight
  Interventions: Diagnostic Test: Neurocognitive, neuromuscular and neurosensitive tests.

INTERVENTIONS:
Diagnostic Test: Neurocognitive, neuromuscular and neurosensitive tests. — At T0, the subject realizes a neurocognive test and an self-assessment of health symptoms autonomously on its professional digital tablet. They also realizes two self questionnaires on their state of fatigue (Samn-Perelli Fatigue Scale) and anxiety (Hospital Anxiety and Depression scale).
  At T0 + 3 months, the subject follows a standardized medical examination carried out by a physician, assessing neuromuscular score using the Medical Research Council questionnaire and assessing neurosensitivity score using the Incat Sensory Sum Score. If necessary, the DN4 questionnaire for neuropathic pain is used. The same neurocognitive tests than T0, and Samn-Perelli Fatigue Scale and Hospital Anxiety and Depression scale are also repeated.

SUMMARY:
The subject of the study focuses on commercial aircraft's cabins air quality, under conditions of both fume events and non-fume events. It also delves into the immediate and delayed repercussions of these events on the health of aviation crew members. The expological facet of this study is directed at the detection and quantification of organophosphorus compounds originating from engine oils. The epidemiological facet is geared towards the identification of potential neurological consequences.

DETAILED DESCRIPTION:
The study has two components, one in the field of expology and the other in epidemiology.

The first part will involve instantaneous atmospheric measurement of organophosphorus additives in oils, namely TCP isomers, TXP isomers (commercially available) and TBP, during any fume event, using a portable device developed for this type of event (pre-positioned on all aircraft), over a short time span (around 1 h).

An identical measurement campaign will be systematically carried out on a "control" flight free of fume event, within a week. The aim of this experiment is to sample all fume event (around 100) occurring over a period of 12 months and as many fume event free flights.

At the same time, carbon monoxide will be measured along with organophosphates during the event.

In parallel with these measurements, a "flight self-questionnaire" will be compiled on flight characteristics and cabin environmental conditions will be completed by the flight's in-charge.

The second epidemiological phase will take place in two stages. Each measurement, whether or not it concerns event or not, will be coupled with a systematic self-questionnaire collection of symptoms experienced during the flight, reported by exposed and non-exposed flight crews.

(T0), no later than 72 hours after the end of the flight.

In addition, in order to identify acute and delayed neurological impairment and to assess cognitive functions, each subject included (exposed and unexposed) will perform :

* A self-assessment within 72 hours (Phase 1) and 3 months later (Phase 2) of their neurocognitive performance using the CANTAB (Cambridge Neuropsychological Test Automated Battery) coupled with a self-assessment of fatigue and anxiety levels using self-questionnaires.
* A medical consultation 3 months later (Phase 2), including a standardized medical check-up with neuromuscular and neurosensory tests, self-questionnaires and neurocognitive evaluation identical to those used in Phase 1.

Phase 2 is carried out three months after exposure, in order to investigate effects with a latency up to 5 weeks after exposure.

ELIGIBILITY:
Inclusion Criteria:

* be of legal age (18 years)
* have signed the consent form

Exclusion Criteria:

* be pregnant
* be over 67 years of age

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy aircrew population of a French airline exposed with (exposed) and whithout (non-exposed) fume events.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive self-assessment tests on digital tablet - CANTAB test battery: Paired Associates Learning | Inclusion and month 3
  Boxes are displayed on the screen and are "opened" in a randomised order. One or more of them will contain a pattern. The patterns are then displayed in the middle of the screen, one at a time and the participant must select the box in which the pattern was originally located.
Neurocognitive self-assessment tests on digital tablet - CANTAB test battery: Rapid Visual Information Processing | Inclusion and month 3
  A white box is shown in the centre of the screen, inside which digits from 2 to 9 appear in a pseudo-random order, at the rate of 100 digits per minute. Participants are requested to detect target sequences of digits. When the participant sees the target sequence they must respond as quickly as possible.
Neurocognitive self-assessment tests on digital tablet - CANTAB test battery: One Touch Stockings of Cambridge | Inclusion and month 3
  The participant is shown two displays containing three coloured balls. The displays are presented in such a way that they can be easily perceived as stacks of coloured balls held in stockings or socks suspended from a beam. This arrangement makes the 3-D concepts involved apparent to the participant and fits with the verbal instructions.
Neurosensitive test to explore superficial and deep sensitivity deficits in peripheral neuropathies | At month 3
  Neurosensitive test performed by the doctor during the medical consultation using the Incat Sensory Sum Score (total score: 0-20 with 0: normal sensitivity and 20: very severe sensitivity deficit; each part of the body is graduated from 0: normal sensitivity to 4: very severe sensitivity deficit).
Neuromuscular test to evaluate muscle strength assessment | At month 3
  Neuromuscular test performed by the doctor during the medical consultation using the Medical Research Council questionnaire (total score: 0-60 with 0:.complete tetraplegia and 60: normal muscle strength; each muscular group to a score ranging 0: no visible contraction and 5: normal muscle strength).
Symptoms experienced during the flight or within 72 hours after the flight, duration of symptoms, symptoms experienced previously outside the flight | Inclusion and month 3
  Collect of symptoms by self-administered questionnaire on professional electronic tablet

SECONDARY OUTCOMES:
Characteristics of plane and fume event and possible causes of fume event | Inclusion
  Characteristics of plane and fume event recorded by a self-administered questionnaire to the Chief Flight Attendant. the information collected is:
  aeroplane type; aerodrome of departure and arrival; meteorological conditions at take-off and landing; characteristics of the occurrence for flights with fume event (phase of flight during the occurrence, estimated duration, nature of the occurrence, location, potential sources of contamination).
Measurement of organophosphorus and carbon monoxide in cabin air using an air sampler and a piston syringe. | Inclusion
  Sampling of flight with and without fume event. A short-term (1h) selected organophosphates measurments after all reported fume event on board, by means of a small air sampler operated by flight crew as well as measurements in a similar flight (control) without fume event is carried out during the following week.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda BENSEFA-COLAS, Study Director — National Institute of Health and Medical Research
Locations (1):
- Air France DP.ZM Service de Santé au travail de Roissy-Charles-de-Gaulle, Roissy CDG, France

IPD SHARING:
Plan to Share IPD: No